CLINICAL TRIAL: NCT04255446
Title: An Observational, Controlled, Single Centre Study Validating the Structured Light Plethysmography Against Standard of Care in the Diagnosis and Monitoring of Dysfunctional Breathing
Brief Title: Structured Light Plethysmography Against Standard of Care in the Diagnosis and Monitoring of Dysfunctional Breathing
Acronym: SLPDB
Status: Not yet recruiting | Type: Observational
Sponsor: Pneumacare Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: PCL-SLPDB-2020
Record Dates: First submitted 2020-01-24; First posted 2020-02-05 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Dysfunctional Breathing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dysfunctional Breathing: Patients with Dysfunctional breathing age between 16 to 75 will be included.
  Interventions: Device: Thora3DiTM
- Healthy Volunteers: Healthy Volunteers without any respiratory problems age between 16 to 75 will be included.
  Interventions: Device: Thora3DiTM

INTERVENTIONS:
Device: Thora3DiTM — Not international

SUMMARY:
This is an observational, controlled, single-centre study to validate the Thora3Di™ against standard practice in patients who are undergoing investigation for disproportionate breathlessness. The core methodology involves capturing of data during a short period of measurement of breathing using SLP.

DETAILED DESCRIPTION:
Cohort A: This study is a pilot study with four study visits (Screening, Baseline, week 13 and week 26) to generate data to characterise the tidal breathing patterns and parameters with Thora3Di™. Subjects will have a screening visit within 0 to 14 days prior to the first study visit. For each study visit, subjects will be seen in the clinical research facility and have two 5-minute SLP measurements (at rest and on exertion). The SLP measurement should be performed prior to standard lung function tests with minimal impact on clinical time and not change to hospital attendance. Also, each visit subjects will be asked to report concomitant medications and adverse events, and fill several questionnaires forms as outlined in the SOAs.

Cohort B: Healthy subjects will have only one visit for this study. After signing the informed consent form, subjects will undergo two 5-minutes SLP measurements (at rest and on exertion).

ELIGIBILITY:
Inclusion Criteria:

* • Cohort A: Any adult who is presenting with controlled disproportionate breathlessness will be considered for inclusion as a diseased subject (with excluded comorbidities as cause of breathlessness e.g. uncontrolled asthma (GINA 2019 guidelines), uncontrolled cardiac disease, ILO).

  * Cohort B: Any adult who is in good respiratory health will be considered for inclusion as a normal in the study.

Exclusion Criteria:

* Subject unable to sit in an upright position for required period

  * Subjects with significant co morbidities (assessed by the clinician at screening only):
  * Chest wall or spinal deformity e.g. scoliosis OSA, Apnoea hypopnoea index > 30 (if known)
  * Any other significant disease or disorder which, in the opinion of the investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participants' ability to participate in the study
  * BMI > 40
  * Height > 194 cm
  * Female participant who is pregnant, lactating or planning pregnancy during the course of the study
  * Inability to consent/comply with trial protocol

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cohort A: Any adult who is presenting with controlled disproportionate breathlessness will be considered for inclusion as a diseased subject (with excluded comorbidities as cause of breathlessness e.g. uncontrolled asthma (GINA 2019 guidelines), uncontrolled cardiac disease, ILO).
  • Cohort B: Any adult who is in good respiratory health will be considered for inclusion as a normal in the study.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Estabilsih expected value and dispersion of Structured Light Phlethysmography in Dysfunctional breathing patients | 26 weeks
  Measure SLP parameters during the course of the treatment : Baseline, Week 13 and Week 26 at rest and at exertion

SECONDARY OUTCOMES:
Establish a relationship between Structured Light Phlethysmography parameters and patient report outcomes addressed. | 26 weeks
  Compare SLP parameters with patient outcome reports (Nijmegen and St George Respiratory Questionnaires and BPAT and BORG scores during the course of the treatment
Establish different SLP parameters between patients with dysfunctional breathing and healthy subjects. | 26 weeks
  Compare the differences in SLP parameters between patients with dysfunctional breathing and healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Aashish Vyas, MD, Principal Investigator — Royal Preston Hospital
Locations (1):
- Pneuma Care Ltd, Ely, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No